CLINICAL TRIAL: NCT02097992
Title: Effect of Roflumilast on Airway Blood Flow as an Expression of Airway Inflammation in COPD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120591; DAL-IT-06 (Other Grant/Funding Number: FOREST)
Record Dates: First submitted 2014-02-13; First posted 2014-03-27 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: COPD
Keywords: COPD; airway blood flow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SD placebo and MD roflumilast then MD placebo (Experimental): Participants will receive placebo (single dose) followed by a 4 week treatment with 500ug roflumilast daily, followed by a 4 week washout period, followed by a 4 week treatment with placebo daily.
  Interventions: Drug: Roflumilast Placebo; Drug: Roflumilast
- SD placebo and MD placebo then MD roflumilast (Experimental): Participants will receive placebo (single dose) followed by a 4 week treatment with placebo daily, followed by a 4 week washout period, followed by a 4 week treatment with 500ug roflumilast daily.
  Interventions: Drug: Roflumilast Placebo; Drug: Roflumilast
- SD roflumilast and MD placebo then MD roflumilast. (Experimental): Participants will receive 500ug roflumilast (single dose) followed by a 4 week treatment with placebo daily, followed by a 4 week washout period, followed by a 4 week treatment with 500ug roflumilast daily.
  Interventions: Drug: Roflumilast Placebo; Drug: Roflumilast
- SD roflumilast and MD roflumilast then MD placebo (Experimental): Participants will receive 500ug roflumilast (single dose) followed by a 4 week treatment with 500ug roflumilast daily, followed by a 4 week washout period, followed by a 4 week treatment with placebo daily
  Interventions: Drug: Roflumilast Placebo; Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast Placebo — Placebo pill
Drug: Roflumilast — 500 Ug ORAL TABLET
  Other Names: Daliresp

SUMMARY:
The objectives of the proposed study are to determine 1) the effect of a single dose of Roflumilast on airway blood flow (Qaw) (study period 1) and 2) the effect of long-term Roflumilast treatment on airway blood flow reactivity delta Qaw)(study period 2) in patients with stable COPD who use ICS regularly.

DETAILED DESCRIPTION:
Participants will be enrolled in the study for three months There will be 6 study days (visits). The patients will be asked to come to the research laboratory in the morning of the study day. They will be instructed to abstain from ingesting alcoholic beverages or using PDE5 inhibitors the night before the study, and from consuming coffee or caffeinated drinks in the morning of the study day because of their potential acute cardiovascular actions. The patients will also be asked not to have a fatty breakfast on the study day to avoid potential effects of fat on the absorption of roflumilast.

The visits will be separated by at least 48 hours. Study period 1: The patients will be randomized into two arms: roflumilast or placebo. Qaw will be measured before and at 15, 30, 60, 120 and 240min in each arm (parallel design) Study period 2: Patients will be randomized to either roflumilast for 4 weeks or placebo for 4 weeks and airway blood flow reactivity will be measured at the end of the treatment period. The patients will then be taken off medication or placebo for 4 weeks and reassigned to the alternate treatment (roflumilast or placebo) for 4 weeks and airway blood flow reactivity will be measured after the this treatment period (cross-over design).

The treatments will be administered in a double-blind randomized design, using active roflumilast and identically appearing roflumilast placebo provided by Forest.

Visit 1

On this visit, a medical history will be obtained from the patients and they will undergo a physical examination and complete pulmonary function testing. If they meet entry criteria, Qaw will be measured before and 15 min after the inhalation of 180 µg albuterol using a spacer (ΔQaw). We have previously shown that vasodilation peaks between 5 and 30 min after inhaling this dose of albuterol in healthy non-smokers; in patients with COPD, who exhibit a vasodilatory response to inhaled albuterol, the peak effects also occur at the same time as in healthy subjects. Since all patients enrolled in the present study will be regular ICS users, we expect that all of them will have a vasodilator response to albuterol as previously shown.

Visit 2

On this day, Qaw will be measured before and at 15, 30, 60,120 and 240 min after the oral administration of either 500µg roflumilast or placebo, blinded to patient and investigator (acute roflumilast effects).

Visit 3

The patients will be given either 500µg roflumilast or placebo (alternate to treatment at visit 2) blinded to patient and investigator. One hour later, Qaw will be measured before and 15 min after the inhalation of 180µg albuterol using a spacer (ΔQaw). Pharmacokinetic studies have shown that the geometric mean plasma concentration of roflumilast after a 500µg dose peaks at one hour after oral drug administration.

The patients will then be randomized in a double blind fashion to either roflumilast 500 µg or placebo every morning before breakfast. They will be asked to return for a follow up visit 4 weeks later (visit 4).

Visit 4

The patients will not take their morning dose (roflumilast or placebo) on this day. Qaw will be measured before and 15 min after the inhalation of 180 µg albuterol using a spacer (ΔQaw). The treatment will be discontinued and the patients will be asked to return for visit 5 after a 4-week washout period.

Visit 5

The protocol of visit 4 will be repeated. The patients will then be started on the alternate treatment for 4 weeks: Those on roflumilast between visits 3 and 4 will now be placed on placebo, and those on placebo between visits 3 and 4 will be placed on roflumilast. The patients will be asked to return for a final visit (visit 6) 4 weeks later.

Visit 6

The protocol of visit 4 will be repeated. The patients will then undergo an exit exam and be discharged from the study

ELIGIBILITY:
Inclusion Criteria:

* Twenty-four patients with physician-diagnosed COPD (female and male, current smokers or ex-smokers) over the age of 45 years will be recruited for this study.
* The patients will have to have a smoking history of at least 10 pack-years, and they must have been using an ICS regularly for at least 4 weeks at the time of screening.
* Confirmation of the diagnosis of COPD will require the presence of persistent exertional dyspnea and a post-bronchodilator FEV1 of less than 80% of predicted and FEV1/FVC ratio less than 0.7 (GOLD stage ≥2). At entry into the study, the patients will have to be clinically stable; they will be allowed to remain on their regular COPD treatment regimen and use a LABA and/or LAMA until 24 hours before, and a SABA and/or short-acting muscarinic antagonist (SAMA) until 6 hours before coming to the laboratory. If using roflumilast, the subjects will have to discontinue it 4 weeks before entering into the study.-

Exclusion Criteria:

* Women of childbearing potential who do not use accepted birth control measures
* Pregnant and breast-feeding women.
* Use of cardiovascular medications that cannot be held on the study days
* Use of oral airway medications or anti-inflammatory agents
* Use of supplemental oxygen that cannot be discontinued during the laboratory visit
* Subjects with known SABA or roflumilast intolerance
* An acute COPD exacerbation within four weeks prior to the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Divison of Pulmonary and Critical Care Medicine, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Treatment 1 (1 Day)
Arm/Group | SD Placebo and MD Roflumilast Then MD Placebo | SD Placebo and MD Placebo Then MD Roflumilast | SD Roflumilast and MD Placebo Then MD Roflumilast. | SD Roflumilast and MD Roflumilast Then MD Placebo
Started | 2 | 3 | 4 | 2
Completed | 2 | 3 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Treatment 2 (4 Weeks)
Arm/Group | SD Placebo and MD Roflumilast Then MD Placebo | SD Placebo and MD Placebo Then MD Roflumilast | SD Roflumilast and MD Placebo Then MD Roflumilast. | SD Roflumilast and MD Roflumilast Then MD Placebo
Started | 2 | 3 | 4 | 2
Completed | 2 | 3 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | SD Placebo and MD Roflumilast Then MD Placebo | SD Placebo and MD Placebo Then MD Roflumilast | SD Roflumilast and MD Placebo Then MD Roflumilast. | SD Roflumilast and MD Roflumilast Then MD Placebo
Started | 2 | 3 | 4 | 2
Completed | 2 | 3 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Treatment 3 (4 Weeks)
Arm/Group | SD Placebo and MD Roflumilast Then MD Placebo | SD Placebo and MD Placebo Then MD Roflumilast | SD Roflumilast and MD Placebo Then MD Roflumilast. | SD Roflumilast and MD Roflumilast Then MD Placebo
Started | 2 | 3 | 4 | 2
Completed | 2 | 3 | 4 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SD Placebo and MD Roflumilast Then MD Placebo | SD Placebo and MD Placebo Then MD Roflumilast | SD Roflumilast and MD Placebo Then MD Roflumilast. | SD Roflumilast and MD Roflumilast Then MD Placebo | Total
Number analyzed (Participants) | 2 | 3 | 4 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4 | 2 | 10
  >=65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 0 | 2
  Male | 2 | 3 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Airway Blood Flow Reactivity (Delta Qaw)
Description: percentage of change on airway blood flow induced by albuterol.
Time Frame: Immediate or 4 weeks
Measure: Mean (Standard Error); unit: % of change
Groups:
- Long Term Multidose Roflumilast or Placebo: Treatment with 500ug roflumilast or placebo for 4 weeks
- Acute Roflumilast or Placebo: Treatment with a single dose of 500ug roflumilast or placebo
Arm/Group | Long Term Multidose Roflumilast or Placebo | Acute Roflumilast or Placebo
Number analyzed (Participants) | 11 | 11
% of change
  roflumilast | 29.1 (6.8) | 13.7 (9.5)
  placebo | 8.9 (4.6) | 15.6 (10.3)

ADVERSE EVENTS:
Groups:
- Single Dose Roflumilast: Participants received a single dose of 500Ug of Roflumilast for one day.
- Single Dose Placebo: Participants received a single dose Placebo for one day.
- Multi-dose Roflumiast: Participants received a daily dose of 500Ug of Roflumilast for four weeks.
- Multi-dose Placebo: Participants received a daily Placebo dose for four weeks
Arm/Group | Single Dose Roflumilast | Single Dose Placebo | Multi-dose Roflumiast | Multi-dose Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 1/11 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose Roflumilast (N=6) | Single Dose Placebo (N=5) | Multi-dose Roflumiast (N=11) | Multi-dose Placebo (N=11)
increase of cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The number of patients enrolled was lower than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No